CLINICAL TRIAL: NCT04181008
Title: Pharmacokinetics of Amiloride Nasal Spray in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Center for Addiction and Mental Health (Unknown)
Responsible Party: Principal Investigator, Venkata Yellepeddi, Associate Professor, Division of Clinical Pharmacology, University of Utah
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 126328
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Amiloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.2 mg (Experimental)
  Interventions: Drug: Amiloride
- 0.4 mg (Experimental)
  Interventions: Drug: Amiloride
- 0.6 mg (Experimental)
  Interventions: Drug: Amiloride

INTERVENTIONS:
Drug: Amiloride — Amiloride Nasal Spray
  Other Names: Midamor
  Arms: 0.2 mg
Drug: Amiloride — Amiloride Nasal Spray
  Other Names: Midamor
  Arms: 0.4 mg
Drug: Amiloride — Amiloride Nasal Spray
  Other Names: Midamor
  Arms: 0.6 mg

SUMMARY:
This study is a single-center, open-label study of the plasma pharmacokinetics of amiloride nasal spray at three different doses in healthy volunteers.

DETAILED DESCRIPTION:
In this clinical study, we will evaluate the plasma pharmacokinetics of amiloride nasal spray in healthy volunteers at three different doses. The data obtained from this study will provide us with pharmacokinetic information that will help develop dosing regimens for future clinical efficacy studies in anxiety patients. Currently, there is no information on the bioavailability and pharmacokinetics of amiloride in humans after intranasal administration. All participants will be allowed to self-administer amiloride nasal spray at 0.2, 0.4, and 0.6 mg doses of amiloride. A series of timed blood samples (0,10, 15, 30, 60 minutes, and 4, 6, 8, 12 and 24 hours,1mL each time point) will be collected.

Primary objectives:

1. To evaluate the pharmacokinetics of amiloride nasal spray at three different doses 0.2, 0.4, and 0.6 mg in healthy human volunteers.
2. To calculate the following pharmacokinetic parameters after intranasal administration of amiloride: time to reach maximum plasma concentration (Tmax), maximum plasma concentration (Cmax), area under the curve (AUC), the volume of distribution (Vd) and clearance (CL).

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 to 30 years of age.
* Females between 18 to 30 years of age.
* Provide written informed consent and authorization.
* Study participants must be able to complete consent, all study evaluations, olfactory testing, and study-related health questionnaires written in the English language.

Exclusion Criteria:

* History of chronic drug, or narcotic abuse.
* Chronic use of tranquilizers, sedatives, aspirin, antibiotics, or other medications.
* Non-English speaking / English translation services required
* Unwilling or unable to provide informed, written consent.
* History or presence of major organ dysfunction.
* History of malignancy, stroke, or diabetes; cardiac, renal, liver, or severe gastrointestinal disease; or other serious illness.
* History of conditions which might contraindicate or require caution be used in the administration of amiloride including hyperkalemia with elevated serum potassium levels (greater than 5.5 mEq per liter), currently receiving other potassium-conserving agents such as spironolactone or triamterene, currently receiving potassium supplementation in the form of medication, potassium-containing salt substitutes or a potassium-rich diet, history or diagnosis of hypersensitivity to Amiloride.
* Subjects with abnormal kidney function tests [estimated glomerular filtration (eGFR) - < 60, and albumin to creatinine ratio (ACR) - > 30]
* Female subjects who are pregnant or nursing at the time of screening.
* Subjects who underwent any kind of surgery of nose and septum within the past one year.
* Subjects diagnosed with chronic rhinosinusitis.
* Treatment with any other investigational drug during the 30 days prior to enrollment into the study.
* Subjects who smoke, have a history of smoking or use nicotine-containing products.
* Subjects who have donated blood within 30 days prior to study entry, including that withdrawn during the conduct of any other clinical study.
* Subjects presenting with acute illness.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
amiloride plasma concentration | 10 minutes
amiloride plasma concentration | 15 minutes
amiloride plasma concentration | 30 minutes
amiloride plasma concentration | 60 minutes
amiloride plasma concentration | 2 hours
amiloride plasma concentration | 4 hours
amiloride plasma concentration | 6 hours
amiloride plasma concentration | 8 hours
amiloride plasma concentration | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Venkata K Yellepeddi, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weissman MM, Klerman GL, Markowitz JS, Ouellette R. Suicidal ideation and suicide attempts in panic disorder and attacks. N Engl J Med. 1989 Nov 2;321(18):1209-14. doi: 10.1056/NEJM198911023211801. PMID 2797086
- [Background] Grant BF, Saha TD, Ruan WJ, Goldstein RB, Chou SP, Jung J, Zhang H, Smith SM, Pickering RP, Huang B, Hasin DS. Epidemiology of DSM-5 Drug Use Disorder: Results From the National Epidemiologic Survey on Alcohol and Related Conditions-III. JAMA Psychiatry. 2016 Jan;73(1):39-47. doi: 10.1001/jamapsychiatry.2015.2132. PMID 26580136
- [Background] Meuret AE, Rosenfield D, Wilhelm FH, Zhou E, Conrad A, Ritz T, Roth WT. Do unexpected panic attacks occur spontaneously? Biol Psychiatry. 2011 Nov 15;70(10):985-91. doi: 10.1016/j.biopsych.2011.05.027. Epub 2011 Jul 23. PMID 21783179
- [Background] Maddock RJ, Buonocore MH, Miller AR, Yoon JH, Soosman SK, Unruh AM. Abnormal activity-dependent brain lactate and glutamate+glutamine responses in panic disorder. Biol Psychiatry. 2013 Jun 1;73(11):1111-9. doi: 10.1016/j.biopsych.2012.12.015. Epub 2013 Jan 17. PMID 23332354
- [Background] Battaglia M, Pesenti-Gritti P, Medland SE, Ogliari A, Tambs K, Spatola CA. A genetically informed study of the association between childhood separation anxiety, sensitivity to CO(2), panic disorder, and the effect of childhood parental loss. Arch Gen Psychiatry. 2009 Jan;66(1):64-71. doi: 10.1001/archgenpsychiatry.2008.513. PMID 19124689
- [Background] Spatola CA, Scaini S, Pesenti-Gritti P, Medland SE, Moruzzi S, Ogliari A, Tambs K, Battaglia M. Gene-environment interactions in panic disorder and CO(2) sensitivity: Effects of events occurring early in life. Am J Med Genet B Neuropsychiatr Genet. 2011 Jan;156B(1):79-88. doi: 10.1002/ajmg.b.31144. Epub 2010 Nov 30. PMID 21184587
- [Background] D'Amato FR, Zanettini C, Lampis V, Coccurello R, Pascucci T, Ventura R, Puglisi-Allegra S, Spatola CA, Pesenti-Gritti P, Oddi D, Moles A, Battaglia M. Unstable maternal environment, separation anxiety, and heightened CO2 sensitivity induced by gene-by-environment interplay. PLoS One. 2011 Apr 8;6(4):e18637. doi: 10.1371/journal.pone.0018637. PMID 21494633
- [Background] Cittaro D, Lampis V, Luchetti A, Coccurello R, Guffanti A, Felsani A, Moles A, Stupka E, D' Amato FR, Battaglia M. Histone Modifications in a Mouse Model of Early Adversities and Panic Disorder: Role for Asic1 and Neurodevelopmental Genes. Sci Rep. 2016 Apr 28;6:25131. doi: 10.1038/srep25131. PMID 27121911
- [Background] Giannese F, Luchetti A, Barbiera G, Lampis V, Zanettini C, Knudsen GP, Scaini S, Lazarevic D, Cittaro D, D'Amato FR, Battaglia M. Conserved DNA Methylation Signatures in Early Maternal Separation and in Twins Discordant for CO2 Sensitivity. Sci Rep. 2018 Feb 2;8(1):2258. doi: 10.1038/s41598-018-20457-3. PMID 29396481
- [Background] Smoller JW, Gallagher PJ, Duncan LE, McGrath LM, Haddad SA, Holmes AJ, Wolf AB, Hilker S, Block SR, Weill S, Young S, Choi EY, Rosenbaum JF, Biederman J, Faraone SV, Roffman JL, Manfro GG, Blaya C, Hirshfeld-Becker DR, Stein MB, Van Ameringen M, Tolin DF, Otto MW, Pollack MH, Simon NM, Buckner RL, Ongur D, Cohen BM. The human ortholog of acid-sensing ion channel gene ASIC1a is associated with panic disorder and amygdala structure and function. Biol Psychiatry. 2014 Dec 1;76(11):902-10. doi: 10.1016/j.biopsych.2013.12.018. Epub 2014 Jan 18. PMID 24529281
- [Background] Battaglia M, Rossignol O, Bachand K, D'Amato FR, De Koninck Y. Amiloride modulation of carbon dioxide hypersensitivity and thermal nociceptive hypersensitivity induced by interference with early maternal environment. J Psychopharmacol. 2019 Jan;33(1):101-108. doi: 10.1177/0269881118784872. Epub 2018 Jul 3. PMID 29968500
- [Background] Chapman CD, Frey WH 2nd, Craft S, Danielyan L, Hallschmid M, Schioth HB, Benedict C. Intranasal treatment of central nervous system dysfunction in humans. Pharm Res. 2013 Oct;30(10):2475-84. doi: 10.1007/s11095-012-0915-1. Epub 2012 Nov 8. PMID 23135822
- [Background] Yellepeddi VK. Stability of extemporaneously prepared preservative-free prochlorperazine nasal spray. Am J Health Syst Pharm. 2018 Jan 1;75(1):e28-e35. doi: 10.2146/ajhp160531. PMID 29273610
- [Background] Knowles MR, Church NL, Waltner WE, Yankaskas JR, Gilligan P, King M, Edwards LJ, Helms RW, Boucher RC. Aerosolized amiloride as treatment of cystic fibrosis lung disease: a pilot study. Adv Exp Med Biol. 1991;290:119-28; discussion 129-32. doi: 10.1007/978-1-4684-5934-0_14. No abstract available. PMID 1950741
- [Background] Knowles MR, Church NL, Waltner WE, Yankaskas JR, Gilligan P, King M, Edwards LJ, Helms RW, Boucher RC. A pilot study of aerosolized amiloride for the treatment of lung disease in cystic fibrosis. N Engl J Med. 1990 Apr 26;322(17):1189-94. doi: 10.1056/NEJM199004263221704. PMID 2157983
- [Background] Noone PG, Regnis JA, Liu X, Brouwer KL, Robinson M, Edwards L, Knowles MR. Airway deposition and clearance and systemic pharmacokinetics of amiloride following aerosolization with an ultrasonic nebulizer to normal airways. Chest. 1997 Nov 5;112(5):1283-90. doi: 10.1378/chest.112.5.1283. PMID 9367469
- [Background] Olivier KN, Bennett WD, Hohneker KW, Zeman KL, Edwards LJ, Boucher RC, Knowles MR. Acute safety and effects on mucociliary clearance of aerosolized uridine 5'-triphosphate +/- amiloride in normal human adults. Am J Respir Crit Care Med. 1996 Jul;154(1):217-23. doi: 10.1164/ajrccm.154.1.8680683.
- [Background] Sood N, Bennett WD, Zeman K, Brown J, Foy C, Boucher RC, Knowles MR. Increasing concentration of inhaled saline with or without amiloride: effect on mucociliary clearance in normal subjects. Am J Respir Crit Care Med. 2003 Jan 15;167(2):158-63. doi: 10.1164/rccm.200204-293OC. Epub 2002 Oct 31. PMID 12411282
- See also: Amiloride Hydrochloride, Drug Label Information — https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=e0cc2d44-436a-47e8-a890-589882fff4c4
- See also: FDA Approval of SPRAVATO™ (esketamine) CIII Nasal Spray for Adults with Treatment-Resistant Depression — https://www.janssen.com/janssen-announces-us-fda-approval-spravato-esketamine-ciii-nasal-spray-adults-treatment-resistant